CLINICAL TRIAL: NCT04475224
Title: A Non-randomized, Multicenter, Confirmatory Study by Intrathecal Administration of KP-100IT in Subjects With Acute Spinal Cord Injury
Brief Title: Phase 3 Study of KP-100IT in Subjects With Acute Spinal Cord Injury
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kringle Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KP-100-ND004
Record Dates: First submitted 2020-07-12; First posted 2020-07-17 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Acute Spinal Cord Injury
Keywords: Hepatocyte Growth Factor; HGF; KP-100IT; KP-100; Intrathecal injection
MeSH Terms: conditions — Deafness, Autosomal Recessive 39 | interventions — Hepatocyte Growth Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label (Other)
  Interventions: Drug: KP-100IT

INTERVENTIONS:
Drug: KP-100IT — Intrathecal injection of 0.6 mg HGF starting at 72 hours since the injury and repeating weekly 5 times
  Other Names: Hepatocyte Growth Factor; HGF

SUMMARY:
This study is non-randomized, multicenter, confirmatory study by intrathecal administration of KP-100IT, code of HGF (Hepatocyte Growth Factor ) formulation for intrathecal injection, in subjects with acute spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* At the time of consent (whether oral or written consent), the patient's age is over 18 years old and under 89 years old
* Patients who have suffered a cervical spinal cord injury within the past 78 hours whose AIS classification was A at 66 - 78 hours after injury-Written informed consent has been obtained

Exclusion Criteria:

* The injury site is C1-C2 or C2-C3
* The patient cannot start rehabilitation necessary for recovery of function at an early stage, for example because tracheal intubation, tracheotomy, or mechanical ventilatory support is necessary
* It is predicted that it will not be possible to administer the first dose of the study drug within 78 hours after the cervical spinal cord injury
* A history of SCI (Spinal cord injury), or abnormal findings in the spinal cavity or marked breakdown of the meninges other than SCI
* Efficacy and safety cannot be evaluated properly due to such as concurrent multiple external trauma or concurrent organ injury
* High dose steroid therapy administered for spinal cord injury
* Disease such as serious liver disorder, renal disease, heart disease, blood dyscrasia, metabolic disease, or infections requiring systemic therapy
* History of malignant tumor
* Participation in a clinical study or research of pharmaceuticals or medical devices within 1 month before registration
* Drug allergies to drugs that will be (or may be) used
* Administration of the study drug to the site of spinal cord injury is inappropriate for a reason such as intrathecal infection or intrathecal mass
* Problems with the subject's ability to give informed consent in person
* The subject is breastfeeding or possibly pregnant
* The subject cannot be expected to survive more than 180 days after the start of administration of the study drug, in the judgement of the investigator
* It is inappropriate for the subject to be included in the study, in the judgement of the investigator

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with an improvement of at least two AIS (American Spinal Injury Association) grade, A to C/D, at 24 weeks after administration | 24 weeks

SECONDARY OUTCOMES:
Time course of ASIA motor score (total/ upper extremity / lower upper extremity) | up to 24weeks
Time course of ASIA sensory score | up to 24weeks
Time course of AIS classification | up to 24weeks
Time course of modified Frankel classification | up to 24weeks
Time course of neurological level of injury | up to 24weeks
Percentage of subjects improving by at least 10 points on the ASIA motor score at 12 weeks and 24 weeks after administration relative to before study drug administration | 12 weeks and 24 weeks
Time courses of plasma concentration and cerebrospinal fluid concentration of KP-100IT after intrathecal administration | up to 24weeks
Evaluation of adverse events | up to 24weeks

CONTACTS AND LOCATIONS:
Overall Officials: Etsuro Hashimura, Study Director — Kringle Pharma, Inc.
Locations (5):
- Japan (5):
  - Spinal Injuries Center, Iizuka, Fukuoka
  - Hokkaido Spinal Cord Injury Center, Bibai, Hokkaido
  - Japanese Red Cross Kobe Hospital, Kobe, Hyōgo
  - Aijinkai Rehabilitation Hospital, Takatsuki, Osaka
  - Murayama Medical Center, Musashimurayama, Tokyo